CLINICAL TRIAL: NCT02305056
Title: Study of Tumor Metabolism by Isotopic Tagging in Patients With High-grade Glioma (CARBONOMIC)
Acronym: CARBONOMIC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARBONOMIC
Record Dates: First submitted 2014-11-20; First posted 2014-12-02 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: High-grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C13 N15 Valine (Experimental): Intervention C13 N15 Valine
  Interventions: Drug: C13 N15 Valine

INTERVENTIONS:
Drug: C13 N15 Valine — C13 N15 Valine administration
  Other Names: CARBONOMIC

SUMMARY:
The purpose of the study is to follow tumoral proteins metabolism by in vivo no radioactive isotopic tagging (carbon 13 and nitrogen 15).

DETAILED DESCRIPTION:
The project aims to study protein turnover in glioblastoma using mass spectrometry after 13C-valine incorporation. This will allow to identify proteins in circulation secreted by tumor which could be diagnostic and pronostic biomarkers in patients With High-grade Glioma.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* patient affiliated to social security or similarly regime
* informed consent form signed
* High-grade Glioma tumor suspicion
* Resective surgery indication
* Hematological assessment :

  * neutrophils > 1500/mm3
  * Platelet > 150 000
  * blood Creatinin normal
  * alkaline Phosphatases and transaminases no more than two times normal
  * Bilirubin < 1.5 times normal

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Precedent complete macroscopic tumor resective surgery
* No valid inclusion criteria
* Intratumoral hemorrhage MRI detected
* Treatment anticoagulant or antisludge treatments
* Active Infections and non controled or medical affection or psychiatric intercurrent non treated
* Evolutive cerebral oedema without corticoid response
* Non controled Epilepsy without antiepileptics response
* Karnofsky score < 40%
* Weight > 100 kg
* No possibility of resective surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Mass spectrometry measurement of C13 labelled proteins | during 30 hours

CONTACTS AND LOCATIONS:
Overall Officials: François BERGER, Pr, Principal Investigator — University Grenoble Hospital
Locations (1):
- CLINATEC, Grenoble, France